CLINICAL TRIAL: NCT03236545
Title: Mechanisms of Vascular Dysfunction in Women: Role of Estradiol
Brief Title: Menopause Effects on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Megan M. Wenner, Assistant Professor, University of Delaware
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 385453-18
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No to Low Endogenous Estrogen (Experimental): PMW and young women (YW) will receive medical study clearance after a detailed physical examination. YW will self-administer subcutaneous injections of the gonadotropin-releasing hormone (GnRH) antagonist, ganirelix acetate (Antagon, 0.25 mg/day in 0.5 ml of normal saline, Organon, Inc., West Orange, New Jersey,) daily to suppress endogenous ovarian hormone production (16, 17, 18). This will begin following a separate medical screening at Reproductive Associates of Delaware 48 hours prior to initiating the hormone intervention to rule out other contraindications prior to beginning the treatment. YW will begin using the antagonist on days 26-28 of their menstrual cycle, and continue daily for 10-12 days. The experimental protocol will be conducted in YW after 3-4 days of using the GnRH antagonist. PMW will complete the experimental protocol prior to use of the 17β-estradiol (E2, 0.1 mg/day patch, Vivelle dot; estradiol patch).
  Interventions: Other: No to Low Endogenous Estrogen
- Estrogen Add-Back (Experimental): Estradiol (E2, 0.1 mg/day patch, Vivelle dot; estradiol patch) will be administered for 7 days to both young and PMW. Young women will use the E2 over the last 7 days of Antagon administration.
  Interventions: Other: No to Low Endogenous Estrogen; Other: Estradiol

INTERVENTIONS:
Other: No to Low Endogenous Estrogen — Ganirelix acetate (Antagon) will be used to prevent endogenous production of ovarian hormones in young women. Ganirelix is derived from native GnRH, and acts by competitively blocking GnRH receptors on the pituitary and subsequent pathways. Thus, administration of the GnRH antagonist (GnRHant) suppresses steroidogenesis, leading to low or undetectable serum estrogen and progesterone concentrations, which occurs within two days of initiation of administration (Oberye, Mannaerts, Huisman & Timmer, 1999; Oberye, Mannaerts, Kleijn, & Timmer, 1999).
Other: Estradiol — Short term estradiol administration elicits changes in vascular function in women, and 0.1mg/day patch is the upper recommended limit for hormone therapy in women (Wenner, Taylor, & Stachenfeld, 2011; Moreau, Hildreth, Meditz, Deane & Kohrt, 2012).
  Other Names: Vivelle dot
  Arms: Estrogen Add-Back

SUMMARY:
The purpose of the study is to identify the independent effect of estradiol (E2) on endothelin-1 (ET-1) mediated vasomotor function in women. The study is the first step in recognizing the impact of ovarian hormones on the mechanisms that regulate vascular function in women to provide a better understanding of the cardiovascular efficacy of hormone therapy.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in women (Roger, Go, Lloyd, Adams, Berry, Brown, et al, 2011). Functional changes in the microvasculature occur with aging and precede atherosclerosis, contributing to CVD (Seals, Jablonski, & Donato, 2011). Furthermore, because of the decline in ovarian hormones during menopause, age-related impairments in endothelial function are exacerbated in postmenopausal women (PMW). However, the safety and efficacy of currently available hormone-based therapies remains controversial (Devi, Sugiguchi, Pederson, Abrassart Glodowski, & Nachtigall, 2013: Miller, Black, Brinton, Budoff, Cedars, Hodis, et al, 2009). Endothelin-1 (ET-1) is a potent vasoconstrictor produced and released by endothelial cells and implicated in the development of atherosclerosis (Best, McKenna, Holmes, & Lerman, 1999; Donato, Gano, Eskurza, Silver, Gates, Jablonski, et al, 2009; Ihling, Szombathy, Bohrmann, Brockhaus, Schaefer, & Loeffler, 2009). ET-1 binds to two receptor subtypes, ET-A and ET-B (Yanagisawa, Kurihara, Kimura, Tomobe, Kobayashi, Mitsui, et al, 1988). While both receptors are located on vascular smooth muscle (VSM) and cause vasoconstriction, ET-B receptors are also located on the endothelium and cause vasodilation (Gomez-Sanchez, Cozza, Foecking, Chiou, & Ferris, 1990; Haynes, 1995; Ishikawa, Ihara, Noguchi, Mase, Mino Saeki, et al, 1994). In women, ET-1 preferentially binds to ET-B receptors compared to ET-A receptors, supporting findings of sex differences in ET-1 receptor responses and suggesting ET-B receptors are under hormonal control (Ergul, Shoemaker, Puett, & Tackett, 1998; Kellogg, Liu, & Pergola, 2001; Stauffer, Westby, Greiner, Van Guilder, & Desouza, 2010). In animal models, estradiol (E2) reduces ET-1 mediated vasoconstriction and increases ET-B receptor mRNA (Pederson, Nielsen, Mortensen, Nilas, & Ottesen, 2008). Thus, low levels of E2 in PMW may contribute to impaired vascular function through an ET-B receptor mechanism. However, the interaction between E2 and ET-1 receptor responses on regulating vascular function in women is currently unknown.

The long-term goal of the laboratory is to understand the impact of ovarian hormones on the mechanisms that regulate vascular function in women to provide a better understanding of the cardiovascular efficacy of hormone therapy. The study is the first step in reaching our goal; the objective of the study is to identify the independent effect of E2 on ET-1 mediated vasomotor function in women. The investigators will measure blood flow responses to local heating in the cutaneous circulation during perfusion of ET-1 receptor antagonists via microdialysis, coupled with measures of intracellular protein and receptor expression on endothelial cells and skin punch biopsies (to assess VSM cells) collected from young and PMW while controlling ovarian hormone exposure. Young women will be tested after suppressing ovarian production of E2 and progesterone with a gonadotropin-releasing hormone antagonist (GnRHant), and again after E2 administration; PMW, who are not using hormone therapy, will be tested before and after E2 admin. The central hypothesis is that declines in E2 impair microvascular vasodilatory function due to cellular changes in ET-B receptor expression on endothelial and VSM cells, and that E2 administration reverses these responses.

ELIGIBILITY:
Inclusion Criteria:

* Young women between 18-35 years of age with regular menstrual cycles
* Postmenopausal women between 50-65 years of age and no more than 10 years past menopause
* Non-smoking
* BMI < 30 kg/m2
* Free from known disease (heart disease, cancer, diabetes)

Exclusion Criteria:

* Current use of hormone therapy or within the past year
* Women using Depo-provera or an intra-uterine device (IUD)
* Pregnant, are planning on becoming pregnant, or are breast- feeding.
* History of stable or unstable angina
* Diabetes
* Neurological disease
* Lung disease
* Kidney or liver disease
* Cancer
* Hysterectomy
* Peripheral vascular disease
* History of blood clots
* Heart disease
* Fibroids
* High blood pressure
* Stroke

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Vascular endothelial function | 3 years
  The capacity of the small and large blood vessels to dilate.

SECONDARY OUTCOMES:
Endothelin receptor expression | 3 years
  Venous endothelial cells and skin punch biopsy will be collected and stained for ET-A and ET-B receptor expression

CONTACTS AND LOCATIONS:
Overall Officials: Megan Wenner, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Information will be available through clinicaltrials.gov database within one year of completion of study.
Time Frame: No later than June 30, 2020
Access Criteria: upon request

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Seals DR, Jablonski KL, Donato AJ. Aging and vascular endothelial function in humans. Clin Sci (Lond). 2011 May;120(9):357-75. doi: 10.1042/CS20100476. PMID 21244363
- [Background] Devi G, Sugiguchi F, Pedersen AT, Abrassart D, Glodowski M, Nachtigall L. Current attitudes on self-use and prescription of hormone therapy among New York City gynaecologists. Menopause Int. 2013 Sep;19(3):121-6. doi: 10.1177/1754045313478941. Epub 2013 May 21. PMID 23761315
- [Background] Miller VM, Black DM, Brinton EA, Budoff MJ, Cedars MI, Hodis HN, Lobo RA, Manson JE, Merriam GR, Naftolin F, Santoro N, Taylor HS, Harman SM. Using basic science to design a clinical trial: baseline characteristics of women enrolled in the Kronos Early Estrogen Prevention Study (KEEPS). J Cardiovasc Transl Res. 2009 Sep;2(3):228-39. doi: 10.1007/s12265-009-9104-y. Epub 2009 May 22. PMID 19668346
- [Background] Best PJ, McKenna CJ, Hasdai D, Holmes DR Jr, Lerman A. Chronic endothelin receptor antagonism preserves coronary endothelial function in experimental hypercholesterolemia. Circulation. 1999 Apr 6;99(13):1747-52. doi: 10.1161/01.cir.99.13.1747. PMID 10190886
- [Background] Donato AJ, Gano LB, Eskurza I, Silver AE, Gates PE, Jablonski K, Seals DR. Vascular endothelial dysfunction with aging: endothelin-1 and endothelial nitric oxide synthase. Am J Physiol Heart Circ Physiol. 2009 Jul;297(1):H425-32. doi: 10.1152/ajpheart.00689.2008. Epub 2009 May 22. PMID 19465546
- [Background] Ihling C, Szombathy T, Bohrmann B, Brockhaus M, Schaefer HE, Loeffler BM. Coexpression of endothelin-converting enzyme-1 and endothelin-1 in different stages of human atherosclerosis. Circulation. 2001 Aug 21;104(8):864-9. doi: 10.1161/hc3301.094742. PMID 11514370
- [Background] Yanagisawa M, Kurihara H, Kimura S, Tomobe Y, Kobayashi M, Mitsui Y, Yazaki Y, Goto K, Masaki T. A novel potent vasoconstrictor peptide produced by vascular endothelial cells. Nature. 1988 Mar 31;332(6163):411-5. doi: 10.1038/332411a0. PMID 2451132
- [Background] Gomez-Sanchez CE, Cozza EN, Foecking MF, Chiou S, Ferris MW. Endothelin receptor subtypes and stimulation of aldosterone secretion. Hypertension. 1990 Jun;15(6 Pt 2):744-7. doi: 10.1161/01.hyp.15.6.744. PMID 2161792
- [Background] Haynes WG. Endothelins as regulators of vascular tone in man. Clin Sci (Lond). 1995 May;88(5):509-17. doi: 10.1042/cs0880509. PMID 7614809
- [Background] Ishikawa K, Ihara M, Noguchi K, Mase T, Mino N, Saeki T, Fukuroda T, Fukami T, Ozaki S, Nagase T, et al. Biochemical and pharmacological profile of a potent and selective endothelin B-receptor antagonist, BQ-788. Proc Natl Acad Sci U S A. 1994 May 24;91(11):4892-6. doi: 10.1073/pnas.91.11.4892. PMID 8197152
- [Background] Ergul A, Shoemaker K, Puett D, Tackett RL. Gender differences in the expression of endothelin receptors in human saphenous veins in vitro. J Pharmacol Exp Ther. 1998 May;285(2):511-7. PMID 9580591
- [Background] Kellogg DL Jr, Liu Y, Pergola PE. Selected contribution: Gender differences in the endothelin-B receptor contribution to basal cutaneous vascular tone in humans. J Appl Physiol (1985). 2001 Nov;91(5):2407-11; discussion 2389-90. doi: 10.1152/jappl.2001.91.5.2407. PMID 11641388
- [Background] Stauffer BL, Westby CM, Greiner JJ, Van Guilder GP, Desouza CA. Sex differences in endothelin-1-mediated vasoconstrictor tone in middle-aged and older adults. Am J Physiol Regul Integr Comp Physiol. 2010 Feb;298(2):R261-5. doi: 10.1152/ajpregu.00626.2009. Epub 2009 Nov 25. PMID 19939973
- [Background] Pedersen SH, Nielsen LB, Mortensen A, Nilas L, Ottesen B. Progestins oppose the effects of estradiol on the endothelin-1 receptor type B in coronary arteries from ovariectomized hyperlipidemic rabbits. Menopause. 2008 May-Jun;15(3):503-10. doi: 10.1097/gme.0b013e318156f803. PMID 18188139
- [Background] Wenner MM, Taylor HS, Stachenfeld NS. Progesterone enhances adrenergic control of skin blood flow in women with high but not low orthostatic tolerance. J Physiol. 2011 Feb 15;589(Pt 4):975-86. doi: 10.1113/jphysiol.2010.194563. Epub 2010 Dec 20. PMID 21173076
- [Background] Wenner MM, Haddadin AS, Taylor HS, Stachenfeld NS. Mechanisms contributing to low orthostatic tolerance in women: the influence of oestradiol. J Physiol. 2013 May 1;591(9):2345-55. doi: 10.1113/jphysiol.2012.247882. Epub 2013 Feb 11. PMID 23401618
- [Background] Wenner MM, Stachenfeld NS. Blood pressure and water regulation: understanding sex hormone effects within and between men and women. J Physiol. 2012 Dec 1;590(23):5949-61. doi: 10.1113/jphysiol.2012.236752. Epub 2012 Oct 1. PMID 23027816
- [Background] Oberye JJ, Mannaerts BM, Huisman JA, Timmer CJ. Pharmacokinetic and pharmacodynamic characteristics of ganirelix (Antagon/Orgalutran). Part II. Dose-proportionality and gonadotropin suppression after multiple doses of ganirelix in healthy female volunteers. Fertil Steril. 1999 Dec;72(6):1006-12. doi: 10.1016/s0015-0282(99)00414-8. PMID 10593372
- [Background] Oberye JJ, Mannaerts BM, Kleijn HJ, Timmer CJ. Pharmacokinetic and pharmacodynamic characteristics of ganirelix (Antagon/Orgalutran). Part I. Absolute bioavailability of 0.25 mg of ganirelix after a single subcutaneous injection in healthy female volunteers. Fertil Steril. 1999 Dec;72(6):1001-5. doi: 10.1016/s0015-0282(99)00413-6. PMID 10593371
- [Background] Stachenfeld NS, DiPietro L, Palter SF, Nadel ER. Estrogen influences osmotic secretion of AVP and body water balance in postmenopausal women. Am J Physiol. 1998 Jan;274(1):R187-95. doi: 10.1152/ajpregu.1998.274.1.R187. PMID 9458917
- [Background] Moreau KL, Hildreth KL, Meditz AL, Deane KD, Kohrt WM. Endothelial function is impaired across the stages of the menopause transition in healthy women. J Clin Endocrinol Metab. 2012 Dec;97(12):4692-700. doi: 10.1210/jc.2012-2244. Epub 2012 Sep 11. PMID 22969140